CLINICAL TRIAL: NCT01424098
Title: A Randomized Controlled Trial of Balance Training in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Balance Training in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roger Goldstein (Other)
Collaborators: Ontario Lung Association (Other)
Responsible Party: Sponsor-Investigator, Roger Goldstein, Director, Respiratory Medicine, West Park Healthcare Centre
Organization: West Park Healthcare Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Goldstein_OTSBalanceRCT_2012
Record Dates: First submitted 2011-08-22; First posted 2011-08-26 (Estimated); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balance Training (Experimental): The treatment group will complete a specific balance training program in addition to conventional pulmonary rehabilitation.
  Interventions: Behavioral: Balance training program
- Usual care (No Intervention): The control group will undergo the usual pulmonary rehabilitation program offered at our centre with no additional balance training classes.

INTERVENTIONS:
Behavioral: Balance training program — Training will consist of 30 minute sessions 3 times/week for 6 weeks in keeping with best practice guidelines for older adults. Sessions will be supervised by physical therapists, using a circuit training approach with different stations designed to target specific areas of impairment. Participants will work through stations in a group setting; however, will receive individualized exercise prescription regarding level of difficulty and exercise progression.
  Arms: Balance Training

SUMMARY:
A growing body of evidence suggests that individuals with chronic lung disease have important deficits in balance control that may be associated with an increased risk of falls. The main purpose of this study is to examine the effects of a balance training program on measures of balance and fall risk in people with chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD; a self-report of decline in balance or fall in the last 5 years or a recent near fall; smoking history greater than 10 pack years; and are able to provide written informed consent.

Exclusion Criteria:

* Inability to communicate because of language skills, hearing or cognitive impairment; and evidence of a neurological or musculoskeletal condition that severely limits mobility and postural control (e.g., cerebrovascular accident, advanced Parkinson's disease, amputation).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | All outcomes will be assessed upon admission to pulmonary rehabilitation (baseline) and again upon completion of the program, an expected average of 6 weeks from baseline.
Balance Evaluation Systems Test | At baseline and 6 weeks.

SECONDARY OUTCOMES:
Balance confidence/falls self-efficacy | At baseline and 6 weeks.
Functional strength | At baseline and 6 weeks.
Self-reported physical function | At baseline and 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Brooks, PhD, Principal Investigator — University of Toronto; Roger S Goldstein, MD, Principal Investigator — West Park Healthcare Centre; Marla K Beauchamp, MSc.PT, Study Chair — University of Toronto; Tania Janaudis-Ferreira, PhD, Study Chair — West Park Healthcare Centre
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Beauchamp MK, Janaudis-Ferreira T, Parreira V, Romano JM, Woon L, Goldstein RS, Brooks D. A randomized controlled trial of balance training during pulmonary rehabilitation for individuals with COPD. Chest. 2013 Dec;144(6):1803-1810. doi: 10.1378/chest.13-1093. PMID 23975185